CLINICAL TRIAL: NCT05540977
Title: Effect of Donepezil on Prevention of Postoperative Urinary Retention in Patients Undergoing Extensive Total Hysterectomy
Brief Title: Donepezil Prevents Urinary Retention After Extensive Total Hysterectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSKY-2022-111-03
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-07

CONDITIONS: Urinary Retention After Procedure
Keywords: Donepezil; Cervical cancer; Urinary Retention
MeSH Terms: conditions — Uterine Cervical Neoplasms; Urinary Retention | interventions — Donepezil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donepezil (Experimental): Patients were randomly divided into experimental group and control group. The experimental group received routine postoperative treatment and took donepezil 5mg orally before going to bed every night from the first day after surgery.
  Interventions: Drug: Donepezil
- Usual care (Other): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Donepezil — Donepezil 5mg QN
  Arms: Donepezil
Other: Usual care — Usual care
  Arms: Usual care

SUMMARY:
Patients were randomly divided into experimental group and control group. The control group received routine postoperative treatment, while the experimental group took donepezil 5mg orally before going to bed every night from the first day after surgery. The catheter was removed and residual urine was measured in both groups 14 days after surgery, the catheter was successfully removed when the residual urine was less than 100ml. After 14 days, the patient was returned to the hospital for residual urine test, and the residual urine was repeated until the residual urine volume was less than or equal to 100ml. The incidence of postoperative urinary retention and adverse drug reactions were compared between the two groups.

DETAILED DESCRIPTION:
This study hypothesized that donepezil could effectively reduce the incidence of urinary retention in cervical cancer patients after extensive total hysterectomy. A total of 108 patients with cervical cancer who underwent abdominal radical hysterectomy in our department from June 1, 2022 to May 31, 2023 were randomly divided into two groups, the experimental group (n = 54) and the control group (n = 54). The incidence of postoperative urinary retention and adverse drug reactions were compared between the two groups.

A. Screening accords with the standard set of subjects, abdominal widely whole palace resection, BiXing random grouping, experimental group from the first day after oral donnelly, pp every night before going to bed together 5 mg, two groups of patients with the rest of the regular place Agreement (including antibiotics to 48 h, postoperative indwelling catheterization, perineum wipe to wash the bid, wound dressing, etc.);

B. The catheter was removed and the residual urine was measured 14 days after operation. The residual urine was ≤100ml, and the catheter was successfully removed. The patients in the experimental group stopped taking the drug, and the residual urine was > 100ml.

C. Residual urine of patients with urinary retention was measured again 14 days later, and the residual urine was ≤100ml. Patients in the experimental group stopped the drug, and the residual urine was > 100ml. Intermittent catheterization was continued, and patients in the experimental group continued to take the drug until the residual urine volume was ≤100ml.

D. This cycle was carried out until the residual urine volume of the last enrolled patient was less than 100ml. The incidence of postoperative urinary retention and adverse drug reactions were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Patients who meet the diagnostic criteria of cervical cancer in the Guidelines for the Diagnosis and Treatment of Cervical Cancer (the Fourth Edition) and have been diagnosed by cervical biopsy or colposcopy
3. Patients with surgical indications undergoing extensive abdominal total hysterectomy
4. The person who signed the informed consent.

Exclusion Criteria:

1. Allergic reaction to donepezil hydrochloride, piperidine derivatives or excipients in preparations
2. Patients with "sick sinus syndrome" or other supraventricular heart conduction diseases
3. Accompanied by serious liver, kidney and other organ dysfunction, serious infectious diseases
4. Patients with a history of mental illness and communication disorders
5. At the time of inclusion, patients with urinary tract infection had a history of urinary tract diseases (stones, congenital malformations, etc.)
6. Patients with intraoperative injury of urinary system, or postoperative ureteral fistula and vesicovaginal fistula.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of urinary retention (residual urine volume < 100ml) | No more than 6 weeks
  Residual urine volume

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No